CLINICAL TRIAL: NCT04484207
Title: Addressing COVID-19 Mental Health Problems Among US Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, Professor of Medical Psychology, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 8006
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Brief Video-based Intervention; Vignette Based Intervention; Non Intervention Control Arm

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video-based intervention (Experimental): A brief video about coping with COVID-19 stress presented to the participants
  Interventions: Other: A short video intervention
- vignette intervention (Experimental): A brief vignette about coping with COVID-19 stress presented to the participants
  Interventions: Other: A vignette intervention
- Control (No Intervention): Only assessment, no intervention arrm

INTERVENTIONS:
Other: A short video intervention — Three minutes video of a veteran that shares his personal story
  Arms: Video-based intervention
Other: A vignette intervention — A written description of the content of the video
  Arms: vignette intervention

SUMMARY:
Coronavirus disease 2019 (COVID-19) has widely and rapidly spread around the world, overwhelming intensive care units and health care capacity. While the physical risk (e.g. pneumonia, respiratory breakdown) is getting the most scientific and clinical attention, this outbreak also has significant mental health risks and extreme psychological fear-related responses. Among the general population, there are high-risk groups as elderly people, disabled individuals and people with previous exposure to trauma (e.g., people with military experience). Veterans are among the subgroups who are high risk for PTSD and other mental health problem. The overarching goal of this study is to examine the efficacy of an online, largescale, brief video-based intervention in reducing fear and stress and improving help seeking behavior in relate to COVID-19.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) has widely and rapidly spread around the world, overwhelming intensive care units and health care capacity, leading the World Health Organization (WHO) to declare a pandemic. According to the official website of the WHO1, more than 3 million people have been confirmed to have a COVID-19 infection, and over than 200,000 deaths have resulted from COVID-19 in almost every area or territories around the world. To effectively cope with the COVID-19 outbreak, various governments have implemented rapid and comprehensive public health emergency interventions that include social restrictions and quarantines, which is the separation and restriction of movement of people who might have been exposed to the virus. Non-essential workers were required to stay at home and the shutdown of non-essential businesses are among the restrictions that influence the lives of millions across the globe. While the physical risk (e.g. pneumonia, respiratory breakdown) is getting the most scientific and clinical attention, this outbreak also has significant mental health risks and extreme psychological fear-related responses.

The outbreak of COVID-19 caused public panic and mental health stress. The rapidly changing information on COVID-19 and the increasing number of confirmed cases and death have elicited fear and anxiety about becoming infected. Isolated at home, people consume information that might be unreliable and unverified for many hours every day. The widespread use of social media and the extensive array (or sources) of information can increase confusion and worries which in turn increases fear and anxiety. Moreover, indirect exposure to 24-hours of television news and social media has a wide range of psychopathological consequences, of which Posttraumatic Stress Disorder (PTSD) symptoms are the most common. A recent study conducted in China one month into the outbreak examined the prevalence of mental health problems in COVID-19 era and found a high rate of depression (48.3%), anxiety (22.6%) and a combination of depression and anxiety (19.4%) among 4,872 people. Furthermore, people with increased social media exposure were almost twice as likely to have depression and anxiety than people with less social media exposure. To date, more than 3 billion people are being asked to stay at home, which may lead to increased exposure to social media, likely resulting in widespread mental health problems among isolated individuals around the globe. Given the magnitude of the COVID-19 outbreak, its risk to physical and mental health,and the unique nature requiring to stay isolated, sheltered, at hospitals, or at home, an effective and timely response is essential to address the psychosocial needs associated with the ongoing exposure to social media, disease, death, and distress.

Among the general population, there are high-risk groups as elderly people, disabled individuals and people with previous exposure to trauma (e.g., people with military experience). Veterans are among the subgroups who are high risk for PTSD and other mental health problem. Furthermore, many veterans are reluctant to seek help, despite enduring symptoms, they avoid mental health care, or may wait years to decades before they seek help. Among reasons to avoid seeking help, patients report mistrust in mental health providers, being seen as weak or stereotyped as "dangerous/violent/crazy", and a belief that they are responsible for having mental health problems. Applying strategies to reduce self-stigma and improve help seeking behavior among veterans may ameliorate impaired functioning and reduce risks for long-term psychiatric illness. Thornicroft showed that social contact is the most effective type of intervention to improve helpseeking behavior and stigma-related attitudes. Social contact involves interpersonal contact with a member of the group; While both direct, in-person social contact and indirect, video-based social contact have effectively improved attitudes toward mental illness, the latter can be implemented on a larger scale. Corrigan and colleagues11 identified the most important ingredients of contact-based programs: an empowered presenter with lived experience who attains his/her goals (e.g., "I was able to fight the COVID-19").

The overarching goal of this study is to examine the efficacy of an online, large-scale, brief video-based intervention in reducing fear and stress and improving help seeking behavior in relate to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* English speakers, veterans (military experience) aged 18-80, US residents

Exclusion Criteria:

* non-English speakers, age less than 18 or more than 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Neria Neria, PhD, Principal Investigator — Columbia University and NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as needed with investigators, IRB etc. A plan will be determined in the short future
Supporting Information: Study Protocol, SAP, ICF
Time Frame: two months
Access Criteria: Co-Is

REFERENCES:
- [Derived] Amsalem D, Lazarov A, Markowitz JC, Gorman D, Dixon LB, Neria Y. Increasing treatment-seeking intentions of US veterans in the Covid-19 era: A randomized controlled trial. Depress Anxiety. 2021 Jun;38(6):639-647. doi: 10.1002/da.23149. Epub 2021 Mar 18. PMID 33734539

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: First, we excluded duplicate submissions, assessments completed in less than minimum expected time, locations (coordinates) outside of the United States, and suspicious IP addresses. Second, we used an open-ended question format requiring the participant's age as a validity question and allowed only a two-digit number as a valid answer and compared responses with age data MTurk provided. Third, we added a question about military trauma with an option of "I did not serve in the military."
Groups:
- Video-based Intervention: A brief video about coping with COVID-19 stress presented to the participants
  A short video intervention: Three minute video of a veteran who shares his personal story
Period: Overall Study
Arm/Group | Video-based Intervention | Vignette Intervention | Control
Started | 86 | 44 | 42
14-Day Follow-Up | 69 | 40 | 33
30-Day Follow-Up | 65 | 34 | 31
Completed | 65 | 34 | 31
Not Completed | 21 | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Video-based Intervention | Vignette Intervention | Control | Total
Number analyzed (Participants) | 86 | 44 | 42 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (14.3) | 45.4 (13.3) | 47.3 (15.6) | 47.2 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 14 | 14 | 54
  Male | 60 | 30 | 28 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 3 | 15
  Not Hispanic or Latino | 79 | 39 | 39 | 157
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 2 | 9 | 23
  White | 64 | 39 | 28 | 131
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 86 | 44 | 42 | 172
Exposure to Military Trauma [Count of Participants; unit: Participants] | 23 | 16 | 10 | 49
Exposure to COVID-19 [Count of Participants; unit: Participants] | 26 | 17 | 17 | 60

OUTCOME MEASURES:

1. Primary Outcome: Help Seeking Intention
Description: Attitudes Toward Seeking Professional Help Scale Minimum value: 3 Maximum value: 12 Higher scores indicate higher help seeking intentions
Time Frame: Assessed at baseline and post-intervention (both day 1), first follow-up (day 14), and second follow-up (day 30)
Population: Using the GEE method, all participants from this arm were analyzed at all time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Video-based Intervention | Vignette Intervention | Control
Number analyzed (Participants) | 86 | 44 | 42
units on a scale
  Baseline | 7.4 (2.7) | 7.9 (2.3) | 7.3 (2.5)
  Post-Intervention | 8.2 (2.5) | 8.1 (2.2) | 7.6 (2.5)
  14-Day Follow-Up | 8.7 (1.1) | 8.7 (1.3) | 8.2 (1.7)
  30-Day Follow-Up | 8.6 (1.2) | 8.6 (1.1) | 8.4 (1.3)
Statistical Analysis 1: Comparison: Video-based Intervention vs Vignette Intervention vs Control; Test type: Superiority; p = 0.031, GEE

2. Secondary Outcome: Help Seeking Intentions Among Veterans Who Reported Anxiety, Depression, or PTSD
Description: Attitudes Toward Seeking Professional Help Scale among veterans who reported anxiety, depression, or PTSD Minimum value: 3 Maximum value: 12 Higher scores indicate higher help seeking intentions
Time Frame: Assessed at baseline and post-intervention (both day 1), first follow-up (day 14), and second follow-up (day 30)
Population: In order to measure this outcome, only veterans from the original sample who reported symptoms of anxiety, depression, or PTSD were analyzed. Using the GEE method, all participants from this arm were analyzed at all time points.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Video-based Intervention: A brief video about coping with COVID-19 stress presented to participants who reported anxiety, depression, or PTSD.
  A short video intervention: Three minute video of a veteran who shares his personal story
- Vignette Intervention: A brief vignette about coping with COVID-19 stress presented to participants who reported anxiety, depression, or PTSD.
  A vignette intervention: A written description of the content of the video
- Control: Only assessment, no intervention arm provided to participants who reported anxiety, depression, or PTSD.
Arm/Group | Video-based Intervention | Vignette Intervention | Control
Number analyzed (Participants) | 54 | 30 | 34
score on a scale
  Baseline | 7.6 [6.9 to 8.3] | 8.1 [7.4 to 8.8] | 7.7 [6.9 to 8.5]
  Post-Intervention | 8.4 [7.9 to 9.1] | 8.1 [7.3 to 8.9] | 8.0 [7.3 to 8.8]
  14-Day Follow-Up | 8.9 [8.3 to 9.6] | 8.5 [8.1 to 9.0] | 8.2 [7.5 to 8.9]
  30-Day Follow-Up | 8.6 [7.9 to 9.3] | 8.3 [7.9 to 8.8] | 8.2 [7.7 to 8.8]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the 30 days of the study period.
Description: Our definitions of adverse event and serious adverse event do not differ from the definitions found on clinicaltrials.gov.
Arm/Group | Video-based Intervention | Vignette Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/44 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/44 | 0/42
Other Adverse Events (participants affected / at risk) | 0/86 | 0/44 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT04484207/Prot_SAP_000.pdf